CLINICAL TRIAL: NCT02914600
Title: A Long-Term Extension Study to Evaluate the Safety of Filgotinib in Subjects With Crohn's Disease
Brief Title: Filgotinib in Long-Term Extension Study of Adults With Crohn's Disease
Acronym: DIVERSITY LTE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: development program for filgotinib for participants with Crohn's disease has been stopped
Sponsor: Galapagos NV (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-419-3896; 2016-002763-34 (EudraCT Number)
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants received blinded treatment during different phases in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Filgotinib 200 mg (Experimental): Participants who received filgotinib 200 milligrams (mg) blinded and completed the parent study, continued to receive filgotinib 200 mg blinded in this study. After unblinding of the parent study, participants continued open-label on filgotinib 200 mg.
  Participants who exited the parent study due to disease worsening or failure to meet response or remission criteria, with the exception of US and Korean males who were not considered dual-biologic refractory, received filgotinib 200 mg open-label in this study.
  Treatment was administered orally once a day until filgotinib becomes commercially available or until the early termination (up to 308 weeks).
  Interventions: Drug: Filgotinib
- Filgotinib 100 mg (Experimental): Participants who received filgotinib 100 mg blinded and completed the parent study, continued to receive filgotinib 100 mg blinded in this study. After unblinding of the parent study, participants continued open-label on filgotinib 100 mg.
  Male participants from the US & Korea who were not considered dual biologic refractory, and who exited the parent study due to disease worsening or failure to meet response or remission criteria, received filgotinib 100 mg open-label in this study.
  Treatment was administered orally once a day until filgotinib becomes commercially available or until the early termination (up to 308 weeks).
  Interventions: Drug: Filgotinib
- Placebo (Placebo Comparator): Participants who received placebo and completed the parent study, continued to receive placebo in this extension study. After unblinding of the parent study, participants on placebo treatment discontinued study drug and study participation.
  Treatment was administered orally once a day until unblinding of the parent study (up to 308 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Filgotinib — Tablet administered orally once a day
  Other Names: GS-6034; GLPG0634; Jyseleca®
  Arms: Filgotinib 100 mg; Filgotinib 200 mg
Drug: Placebo — Tablet administered orally once a day
  Arms: Placebo

SUMMARY:
The primary objective of this study is to observe the long-term safety of filgotinib in adults who have completed or met protocol specified efficacy discontinuation criteria in a prior filgotinib treatment study in Crohn's disease (CD).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of study procedures associated with this trial
* Must have enrolled in a CD parent protocol, GS-US-419-4015, GS-US-419-4016 or GS-US-419-3895 or any other Gilead/Galapagos sponsored filgotinib treatment study for CD
* Females of childbearing potential must have a negative pregnancy test at Day 1 and must agree to continued monthly pregnancy testing during use of filgotinib treatment
* Female participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception for the duration described in the protocol
* Willingness to refrain from live or attenuated vaccines during the study and for 12 weeks after last dose of study drug
* Must have completed all required procedures or met protocol specified efficacy discontinuation criteria in a prior filgotinib treatment study for CD

Key Exclusion Criteria:

* Known hypersensitivity to the study drug
* Any chronic medical condition (including, but not limited to, cardiac or pulmonary disease, alcohol or drug abuse) that, in the opinion of the Investigator or sponsor, would make the individual unsuitable for the study or would prevent compliance with the study protocol
* Females of reproductive potential who are unwilling to abide by protocol-specified contraceptive methods as defined in the protocol
* Use of prohibited concomitant medications as outlined in the study protocol

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1188 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (485):
- United States (100):
  - Digestive Health Specialists Of The Southeast, Dothan, Alabama
  - Arizona Digestive Health - Sun City, Sun City, Arizona
  - Southern California Research Center, Inc., Coronado, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - UC San Diego Health Systems, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - Clearview Medical Research, LLC, Santa Clarita, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - South Denver Gastroenterology, PC, Lone Tree, Colorado
  - Connecticut GI, PC - Research Division, Farmington, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Advanced Research, LLC, Coral Springs, Florida
  - UF Clinical Research Center, Gainesville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida
  - Gulf Region Clinical Research Institute, Pensacola, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Tampa General Hospital, Tampa, Florida
  - Florida Medical Clinic, P.A, Zephyrhills, Florida
  - Gastroenterology Associates Of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Atlanta Gastroenterology Specialist, PC, Suwanee, Georgia
  - Illinois Gastroenterology Group - Arlington Heights, Arlington Heights, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The University of Chicago Medical Center (Clinic), Chicago, Illinois
  - Illinois Gastroenterology Group - Gurnee, Gurnee, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Clinical Trials Unit, Louisville, Kentucky
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital - Crohn's and Colitis Center, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinical Research Center, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - NY Scientific, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - New York University School of Medicine / NYU Gastroenterology Associates, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Carolina's GI Research LLC, Raleigh, North Carolina
  - Fargo Gastroenterology and Hepatology Clinic, Fargo, North Dakota
  - Consultants for Clinical Research, Cincinnati, Ohio
  - UC Health Physicians Clifton, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Options Health Research LLC, Tulsa, Oklahoma
  - Great Lakes Medical Research, LLC, Harrisburg, Pennsylvania
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Vanderbilt University Medical Center - IBD Clinic, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - San Antonio Military Medical Center,, Fort Sam Houston, Texas
  - DHAT Research Institute, Garland, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Baylor College of Medicine - McNair Campus, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Gulf Coast Research Group, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - TDDC San Marcos, San Marcos, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Spring Gastroenterology, The Woodlands, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - HP Clinical Research, Bountiful, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, a division of GI Associates, LLC, Milwaukee, Wisconsin
- Fundacion Estudios Clinicos CiRec, Rosario, Argentina
- Australia (16):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Coastal Digestive Health, Mountain Creek, Queensland
  - Coral Sea Clinical Research Institute (Mackay), North Mackay, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Emeritus Research, Camberwell, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (3):
  - Universitatsklinik Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Abt. Für Inn. Med. & Gastroenterol, (IMuG), Hepatol., Endokrinol., Rheumatol., & Nephrol., Klagenfurt
  - AKH-Medizinische Universitat Wien, Vienna
- Belgium (9):
  - GZA Ziekenhuizen, campus Sint-Vincentius, Antwerp
  - Imelda General Hospital, Bonheiden
  - CUB Hopital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Chretien (CHC) - Clinique Saint-Joseph, Liège
  - CHR Citadelle, Liège
  - AZ Delta, Roeselare
- Bulgaria (4):
  - Medical Center - Complete Medical Solutions OOD, Samokov
  - Medical Center - "Tsaritsa Yoanna" EOOD, Sliven
  - "MDHAT Dr. St.Cherkezov" AD, Veliko Tarnovo
  - MHAT "Sveta Petka" AD, Vidin
- Canada (11):
  - Barrie GI Associates, Barrie
  - University of Calgary, Heritage Medical Research Clinic, Calgary
  - Hamilton Health Sciences Corporation, McMaster University Medical Centre, Hamilton
  - London Health Sciences Centre - University Hospital, London
  - TIDHI Innovation, Inc., North York
  - ABP Research Services, Oakville
  - Royal University Hospital, Saskatoon
  - Mount Sinai Hospital, Toronto
  - The Gordon and Leslie Diamond Health Care Centre, Vancouver
  - Toronto Digestive Disease Associates Inc., Vaughan
  - Percuro Clinical Research Ltd., Victoria
- Croatia (3):
  - University Hospital Center Osijek, Osijek
  - Clinical Hospital Dubrava, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (5):
  - Hepato-Gastroenterology HK, s.r.o., Hradec Králové
  - Oblastni nemocnice Mlada Boleslav, a.s., nemocnice Stredoceskeho kraje, Gastroenterologicke oddeleni, Mladá Boleslav
  - G.E.P. Clinic, s r.o., Prague
  - Thomayerova nemocnice, Interni klinika 3. LF UK a TN, Prague
  - ISCARE a.s. (Klinicke centrum ISCARE), Klinicke a vyzkumne centrum pro strevni zancty, Prague
- France (23):
  - CHU Amiens Picardie, Amiens
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand - Hopital d'Estaing, Clermont-Ferrand
  - APHP - Hopital Beaujon - Clichy - Universite Paris VII, Clichy
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - CHU de Dijon Bourgogne - Hopital Francois Mitterand, Dijon
  - CHU Grenoble Alpes, La Tronche
  - Hopital Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Hopital Nord, Marseille
  - Hopital Saint Joseph, Marseille
  - CHU de Montpellier-Hopital Saint Eloi, Montpellier
  - CHU Hotel-Dieu, Nantes
  - Hopital de l'Archet 2, Nice
  - CHU de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Lyon Sud, Pierre-Bénite
  - CH Annecy Genevois - Site d'Annecy, Pringy
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - CHU de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Nouvel Hopital Civil, Strasbourg
  - Hopitaux Universitaires de Strasbourg - Hopital de Hautepierre, Strasbourg
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - CHU de Nancy - Hopital Brabois Adultes, Vandœuvre-lès-Nancy
- Georgia (3):
  - Unimed Ajara LLC - Batumi Referral Hospital, Batumi
  - Medi Club Georgia LLC, Tbilisi
  - Ltd. Unimed Kakheti - Telavi Referral Hospital, Telavi
- Germany (25):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Medizinisches Versorgungszentrum Delitzsch, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - DRK Kliniken Berlin - Westend - Klinik fuer Innere Medizin, Berlin
  - Stadtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitaetsklinik Koln, Cologne
  - Universitatsklinikum Dresden, Dresden
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - CED Studien UG, Interdisciplinary Crohn Colitis Center (iCCC), Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Westklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Praxis fur Gastroenterologie, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - EUGASTRO GmbH, Leipzig
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum Luneburg, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum der Universitat Munchen - Grosshadern, München
  - Universitaetsmedizin Rostock, Zentrum fuer Innere Medizin, Rostock
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitatsklinikum Ulm, Zentrum Fur Innere Medizin, Ulm
- Greece (5):
  - Hippokration Hospital of Athens, Athens
  - University General Hospital "Attikon", 2nd Propaedeutic Internal Medicine Dept. and Research Unit, Hepatogastroenterology Unit, Athens
  - University General Hospital of Ioannina, Gastroenterology Department, Internal Medicine Division, Ioannina
  - University General Hospital of Patras "Panagia I Voithia", Gastroenterology Department, Internal Medicine Division, Pátrai
  - Hippokratio General Hospital of Thessaloniki "Hippokratio" 4th Internal Medicine Department of Aristotle University of Thessaloniki, Thessaloniki
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Department of Medicine & Therapeutics, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin
  - Tuen Mun Hospital, Tuenmen
- Hungary (8):
  - Bekes Megyei Kosponti Korhaz, Dr. Rethy Pal Tagkorhaz, IV. Belgyogyaszat - 2. Gasztroenterologia, Békéscsaba
  - Szent Margit Korhaz, Gasztroenterológiai Osztály, Budapest
  - Clinexpert Egeszsegugyi Szolgaltato es Kereskedelmi Kft., Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Kozponti Felnott Szakrendelo, Budapest
  - Szent Janos Korhaz es Eszak-budai Egitett Korhazak, I. Belgyogyaszati - Gasztroenterologiai Osztaly, Budapest
  - Debreceni Egyetem Klinikai Kozpont, II. sz. Belgyogyaszati Klinika, Gasztroenterologia, Debrecen
  - Bugat Pal Korhaz, Belgyogyaszat, Gyöngyös
  - Karolina Korhaz es Rendelointezet, Altalanos Belgyogyaszat-Gasztroenterologia, Mosonmagyaróvár
- Landspitali University Hospital, Reykjavik, Iceland
- India (33):
  - Lakeshore Hospital and Research Centre Ltd, Kochi, Kerala
  - Kaizen Hospital, Ahmedabad
  - Victoria Hospital, Bangalore Medical College and Research Institute (BMCRI), Bangalore
  - M S Ramaiah Medical College and Hospital, Bangalore
  - Apollo Speciality Hospital, Chennai
  - VGM Hospital Institute of Gastroenterology, Coimbatore
  - Lourdes Hospital, Ernākulam
  - Fortis Memorial Research Institute, Gūrgaon
  - Gleneagles Global Hospital, Hyderabad
  - Citizens Specialty Hospital, Hyderabad
  - Centre for Liver Research & Diagnostics, Hyderabad
  - SR Kalla Memorial Gastro and General Hospital, Jaipur
  - S.M.S Hospital, Jaipur
  - School of Digestive & Liver Diseases, Kolkata
  - King George's Medical University, Lucknow
  - Dayanand Medical College & Hospital, Ludhiana
  - Kasturba Medical College (KMC) Hospital, Mangaluru
  - Seth G.S. Medical College & KEM Hospital, Mumbai
  - S.L. Raheja Hospital (A Fortis Associate), Mumbai
  - Lokmanya Tilak Municipal General Hospital, Mumbai
  - Midas Multispeciality Hospital Pvt. Ltd, Nagpur
  - Suretech Hospital & Research Centre Ltd, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Department of Surgery, B.J. Government Medical College & Sassoon General Hospital, Pune
  - Grant Medical Foundation Ruby Hall Clinic, Pune
  - Universal Hospital, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Gandhi Hospital, Secunderabad
  - Institute of Gastroenterology & Liver Disease. Sunshine Hospitals, Secunderabad
  - Surat Institute of Digestive Sciences, Surat
  - Kasturba Hospital Medical College, Udupi
  - Sterling Hospital, Vadodara
  - Samvedna Hospital, Varanasi
- Ireland (4):
  - St. Vincent's University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Wellcome Trust HRB Clinical Research Facility, Dublin
  - University Hospital Galway, Galway
- Israel (11):
  - Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Health Care Campus, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir MC, Kefar Sava
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (14):
  - UOC Gastroenterologia II, Castellana Grotte
  - U.O. Fisiopatologia Digestiva, Catanzaro
  - UOC Medicina Interna, Cento
  - Ospedale Clinicizzato SS. Annunziata - Dipartimento di Medicina, Chieti
  - Gastroenterologia clinica - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Endocsopia Digestiva Centralizzata, Milan
  - UO Gastroenterologia, Modena
  - UOC Gastroenterologia, Padua
  - Azienda Ospedaliero-Universitaria Pisana - Presidio Ospedaliero Cisanello, Pisa
  - UOC Gastroenterologia ed Endoscopia Digestiva, Roma
  - UOC di Gastroenterologia ed Endoscopia Digestiva, Roma
  - UOC Medicina Interna a Gastroenterologia, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.S.O. Ordine Mauriziano Di Torino S.C., Torino
- Japan (40):
  - Ohmori Toshihide gastro-intestinal Clinic, Ageo-shi
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital, Chūōku
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Tokai University Hachioji Hospital, Hachiōji
  - Hiroshima Prefectural Hospital, Hiroshima
  - Fukuoka University Hospital, Jonan-ku
  - Saitama Medical Center, Saitama Medical University, Kawagoe
  - Kitakyushu City Hospital Organization Kitakyushu Municipal Medical Center, Kitakyushu-shi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kurume University Hospital, Kurume-shi
  - Hidaka Coloproctology Clinic, Kurume-shi
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - The Jikei University Hospital, Minatoku
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka-shi
  - Iwate Medical University Hospital, Morioka
  - Aichi Medical University Hospital, Nagakute-shi
  - Nagasaki University Hospital, Nagasaki
  - Nagoya City University Hospital, Nagoya
  - Saiseikai Niigata Daini Hospital, Nishiku
  - Hyogo College of Medicine College Hospital, Nishinomiya
  - Okayama University Hospital, Okayama
  - Kinshukai Infusion Clinic, Osaka
  - Osaka City University Hospital, Osaka
  - Wakakusa-Daiichi Hospital, Osaka
  - Ishida IBD Clinic, Ōita
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saga-Ken Medical Centre Koseikan, Saga
  - Saga University Hospital, Saga
  - Tokito Clinic, Saitama
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - National Hospital Organization Sendai Medical Center, Sendai
  - Osaka University Hospital, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - Ieda Hospital, Toyota-shi
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama Health Medicine Association Kannai Suzuki Clinic, Yokohama
- Malaysia (5):
  - Universiti Kebangsaan Malaysia Medical Center, Cheras
  - Hospital Pulau Pinang, George Town
  - Hospital Queen Elizabeth, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
- Netherlands (9):
  - NZW Alkmaar (Noordwest Ziekenhuisgroep), Alkmaar
  - VU Medisch Centrum, Amsterdam
  - Academic Medical Center (AMC), Amsterdam
  - Gelre Hospital, Apeldoorn
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht University Medical Centre, Maastricht
  - Erasmus University Medical Center, Rotterdam
  - Elisabeth-TweeSteden Hospital, Tilburg
  - University Medical Center Utrecht, Utrecht
- New Zealand (7):
  - Christchurch Hospital, Christchurch
  - Southern District Health Board - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Newtown
  - Bay of Plenty District Health Board - Tauranga Hospital, Tauranga
  - Hutt Valley District Health Board - Hutt Valley Hospital, Wellington
- Poland (24):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Klinika Gastroenterologii i Chorob Wewnetrznych, Bialystok
  - VITAMED Galaj i Cichomski spólka jawna, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im. Dr. Jana Biziela w Bydgoszczy, Centrum Endoskopii Zabiegowej, Poradnia Chorob Jelitowych, Bydgoszcz
  - Gabinet Lekarski Janusz Rudzinski, Bydgoszcz
  - NZOZ INTER-MED, Centrum Endoskopowe, Częstochowa
  - Niepubliczny Zaklad Opieki Zdrowotnej ALL-MEDICUS, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Uniwerstyeckiego Szpitala Klinicznego nr 1 im. Norberta Barlickiego, Lodz
  - Trialmed Crs, Piotrkow Trybunalski
  - Clinical Research Center Sp. z o.o. Medic-R Sp.k., Poznan
  - Gabinet Lekarski Dr. Hab. N. Med. Bartosz Korczowski, Rzeszów
  - Endoskopia Sp. z o.o., Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - GASTROMED Kopon, Zmudzkinski i Wspolnicy Sp. j. Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - H-T.Centrum Medyczne Spolka z Ograniczona Odpowiedzialnoscia Sp.K., Tychy
  - Centrum Zdrowia MDM, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administacji w Warszawie, Warsaw
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw
  - Niepubliczny Zaklad Opieki Zrodotnej VIVAMED Jadwige Miecz, Warsaw
  - Bodyclinic, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (8):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitario de Coimbra, E.P.E., Coimbra
  - Centro Hospitalar Cova de Beira, EPE, Covilha
  - Centro Hospitalar do Algarve EPE, Faro
  - Hospital da Senhora da Oliveira Guimaraes, E.P.E., Guimarães
  - Hospital Beatriz Angelo, Loures
  - Centro Hospitalar de Sao Joao, EPE, Porto
  - Unidade Local de Saúde do Alto Minho, Viana do Castelo
- Romania (10):
  - MedLife, Gastroenterologie, Bucharest
  - Spitalul Universitar de Urgenta Militar Central Dr. Carol Davila - Sectia Clinica de Gastroenterologie, Bucharest
  - S.C. Centrul Medical Sana S.R.L., Gastroenterologie, Bucharest
  - Delta Health Care/ Ponderas Academic Hospital, Bucharest
  - Spitalul Clinic Colentina - Sectia de Spitulal Clinic Colentina, Gastroenterologie, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti - Sectia Medicina Interna II, Bucharest
  - Gastromedica SRL, Gastroenterologie, Iași
  - Cabinet Particular Policlinic Algomed SRL, Timișoara
  - Centrul Medical Tuculanu, Gastroenterologie, Timișoara
  - S.C. Policlinica Dr. Citu S.R.L.- Gastroenterologie, Timișoara
- Russia (10):
  - State Budgetary Healthcare Institution "Chelyabinski Regional Clinical Hospital", Chelyabinsk
  - State Budgetary Institution of Health Irkustsk Order "Badge of Honor" Regional Clinical Hospital, Irkutsk
  - State Budgetary Healthcare Institution of Moscow Region "Moscow Regional Clinical Research Institute n.a. M.F. Vladimirskiy", Moscow
  - State Budgetary Healthcare Institution of Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital n.a. N.A., Nizhny Novgorod
  - State Budgetary Healthcare Institution of the Novosibirsk Region "State Novosibirsk Regional Clinical Hospital", Novosibirsk
  - State Budgetary Institution of Health of Novosibirsk Region "City Clinical Hospital #12", Novosibirsk
  - Saint Petersburg State Budgetary Healthcare Institution "City Polyclinic #38", Saint Petersburg
  - "Scientific Research Centre ECO-safety" LLC, Saint Petersburg
  - "PolyClinic EXPERT" LLC, Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
- Serbia (5):
  - Clinical Hospital Center Zemun, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Clinical Center of Serbia, Belgrade
  - Zvezdara University Medical Center, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- Slovakia (3):
  - Cliniq s. r. o., Gastroenterologicke centrum Ruzinov, Bratislava
  - KM Management, s.r.o., Gastroenterologicke a hepatologicke centrum Nitra, Nitra
  - Gastro I., s.r.o., Prešov
- South Africa (3):
  - Dr MJ Prins, Cape Town
  - Dr John P Wright, Cape Town
  - Peermed Clinical Trial Centre, Johannesburg
- South Korea (12):
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Guri-si
  - Hanyang University Guri Hospital, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Division of Gastroenterology, Department of Medicine, Samsung Medical Center, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (13):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Centro Medico Teknon, Barcelona
  - Hospital del Mar, Barcelona
  - Complejo Hospitalario Universitario de Ferrol, Ferrol
  - Hospital Universitario de Gran Canaria "Dr. Negrin", Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital de Montecelo, Pontevedra
  - Hospital de Sagunto, Sagunto
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital de Galdakao-Usandolo, Usansolo
- Sri Lanka (4):
  - National Hospital of Sri Lanka, Colombo
  - Karapitiya Teaching Hospital, Galle
  - Kandy Teaching Hospital, Kandy
  - Colombo North Teaching Hospital, Ragama
- Sweden (2):
  - Danderyds Sjukhus AB, Danderyd
  - Akademiska Sjukhuset, Uppsala
- Switzerland (2):
  - Intesto Gastroenterologische Praxis & Crohn-Colitis-Zentrum Bern, Bern
  - Universitätsspital Zürich, Zurich
- Taiwan (11):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Chang Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation, Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District
- Ukraine (16):
  - Multispecialty Clinical Hospital of Intensive Treatments and Emergency Medical Care, Chernivtsi
  - Regional Municipal Institution "Chernivtsi Regional Clinical Hospital", Surgical Department, Chernivtsi
  - State Institution "Institute of Gastroenterology of National Academy of Medical Sciences of Ukraine", Dnipropetrovsk
  - Ivanto-Frankivsk Central City Clinic Hospital, Therapy Department #1. State Higher Education Institution Ivano-Frankivsk National, Ivano-Frankivsk
  - Municipal Health Care Institution "Kharkiv City Clinical Hospital #2 named after prof. O. O. Shalimov", Proctology Department, Kharkiv
  - Municipal Institution of Health Care "Regional Hospital of War Veterans", Therapeutic Department No1, Kharkiv
  - Treatment and Diagnostic Center of Private Enterprise of Private Production Company "Acinus", Kropyvnytskyi
  - Kyiv City Clinical Hospital No. 18, Proctology Department, Kyiv
  - Municipal Non-profit Enterprise "Consultative and Diagnostic Center" of Pechersk District of Kyiv, Therapy Department, Kyiv
  - Municipal Institution "Odesa Regional Clinical Hospital", Regional Gastroenterology Center based on Surgery Department, Odesa
  - Ternopil Regional Clinical Hospital, Regional Center of Gastroenterology with Hepatology, Ternopil
  - Municipal Institution "Uzhgorod District Hospital", Therapy Department, Uzhhorod
  - Vinnytsia Regional Clinical Hospital of War Veterans, Therapy Department #1, Vinnytsia
  - M.I. Pyrogov Vinnytsia Regional Clinical Hospital, Gastroenterology Department, Vinnytsia
  - Medical Center LLC "Health Clinic", Vinnytsia
  - Municipal Institution "Zaporizhzhya Regional Clinical Hospital" of Zaporizhzhya Regional Council, Zaporizhzhya
- United Kingdom (14):
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich, Norfolk
  - Queen Elizabeth Hospital, Birmingham
  - The Pennine Acute Hospitals NHS Trust, Bury
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Lothian, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Glasgow Clinical Research Facility - Queen Elizabeth University Hospital, Glasgow
  - NHS Greater Glasgow and Clyde, Glasgow
  - Wycombe Hospital, High Wycombe
  - St George's University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, St Mary's Hospital, London
  - Oxford University Hospitals NHS Trust, Oxford
  - St Helens and Knowsley Teaching Hospitals NHS Trust, Prescot
  - Southampton National Institute for Health Research, Wellcome Trust Clinical Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in 37 countries: Australia, Austria, Belgium, Canada, Croatia, Czech Republic, France, Georgia, Germany, Greece, Hong Kong, Hungary, India, Ireland, Israel, Italy, Japan, Malaysia, the Netherlands, New-Zealand, Poland, Portugal, Republic of Korea, Romania, Russia, Serbia, Singapore, Slovakia, South-Africa, Spain, Sri Lanka, Sweden, Switzerland, Taiwan, Ukraine, the United Kingdom, and the United States (US).
Pre-assignment Details: Participants with Crohn's disease (CD), who had completed or met protocol-specified efficacy discontinuation criteria from previous parent studies (GS-US-419-4015 [NCT03046056], GS-US-419-4016 [NCT03077412] or GS-US-419-3895 [GLPG0634-CL-309] [NCT02914561]) were rolled-over to this long-term extension study.
  Sponsor decided not to pursue extension of filgotinib indication for CD, as GS-US-419-3895 did not meet the co-primary endpoint and decided to terminate this study prematurely.
Period: Overall Study
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Started | 945 | 119 | 124
Treated | 944 | 119 | 124
Completed | 0 | 0 | 0
Not Completed | 945 | 119 | 124
Not completed — Adverse Event | 298 | 35 | 25
Not completed — Sponsors decision | 287 | 41 | 12
Not completed — Withdrawal by Subject | 158 | 20 | 18
Not completed — Investigators discretion | 169 | 14 | 13
Not completed — Lost to Follow-up | 10 | 4 | 0
Not completed — Pregnancy | 8 | 0 | 0
Not completed — Protocol Violation | 5 | 3 | 0
Not completed — Non-compliance with study drug | 6 | 1 | 0
Not completed — Death | 3 | 1 | 1
Not completed — Current Study Unblinded and participant confirmed on Placebo | 0 | 0 | 55
Not completed — Enrolled but not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who took at least 1 dose of study drug in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo | Total
Number analyzed (Participants) | 944 | 119 | 124 | 1187
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13.60) | 47 (13.28) | 42 (12.42) | 40 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 514 | 33 | 56 | 603
  Male | 430 | 86 | 68 | 584
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 5 | 0 | 23
  Not Hispanic or Latino | 904 | 112 | 123 | 1139
  Unknown or Not Reported | 22 | 2 | 1 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 137 | 18 | 23 | 178
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 18 | 10 | 3 | 31
  White | 739 | 89 | 96 | 924
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 47 | 2 | 2 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study drug, and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug whether or not considered related to the study drug. Treatment-emergent adverse events (TEAEs) were defined as 1 or both of the following:
  * Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
  * Any AEs leading to premature discontinuation of study drug.
Time Frame: From the First Dose to Week 312
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 944 | 119 | 124
Participants | 820 | 103 | 96

2. Secondary Outcome: Change From Baseline in Patient Reported Outcomes 2 (PRO2) Scores for Liquid or Very Soft Stools
Description: The PRO2 was a composite score based on 2 components of CDAI, the number of liquid or soft stools/day for 7 days, stool frequency and abdominal pain (rated on a scale of 0-3, higher values mean greater abdominal pain) assessed for 7 days. The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The sub scores of abdominal pain (0-3), general well-being (0-4, higher values mean worse well-being), and number of liquid or very soft stools were summed over the 7 days prior to each visit. The remaining predictors were also weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome. Change from baseline for number of liquid or very soft stool per day was reported.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 96, Week 156, Week 216, Week 264, and Week 300
Population: Participants from safety analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Number of liquid/very soft stools/day
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 911 | 113 | 113
Number of liquid/very soft stools/day
  Baseline | 5.6 (3.26) | 4.0 (3.12) | 2.2 (1.92)
  Change at Week 12: number analyzed (Participants) | 787 | 103 | 103
  Change at Week 12 | -1.6 (2.71) | -0.7 (2.01) | 0.2 (1.44)
  Change at Week 24: number analyzed (Participants) | 682 | 89 | 89
  Change at Week 24 | -1.8 (2.89) | -0.7 (2.59) | 0.1 (1.15)
  Change at Week 48: number analyzed (Participants) | 516 | 74 | 81
  Change at Week 48 | -2.0 (3.14) | -0.8 (2.49) | 0.0 (1.21)
  Change at Week 96: number analyzed (Participants) | 305 | 49 | 53
  Change at Week 96 | -2.2 (3.11) | -0.7 (2.70) | 0.4 (2.79)
  Change at Week 156: number analyzed (Participants) | 177 | 30 | 26
  Change at Week 156 | -2.4 (3.14) | -0.7 (3.19) | -0.2 (1.63)
  Change at Week 216: number analyzed (Participants) | 82 | 13 | 6
  Change at Week 216 | -2.8 (3.17) | -1.2 (4.10) | 1.0 (1.41)
  Change at Week 264: number analyzed (Participants) | 20 | 4 | 0
  Change at Week 264 | -2.0 (2.86) | -4.8 (6.18) |
  Change at Week 300: number analyzed (Participants) | 4 | 0 | 0
  Change at Week 300 | 0.0 (2.71) |  |

3. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (PRO2) Scores for Abdominal Pain
Description: The PRO2 was a composite score based on 2 components of CDAI, the number of liquid or soft stools/day for 7 days, stool frequency and abdominal pain (rated on a scale of 0-3, higher values mean greater abdominal pain) assessed for 7 days. The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The sub scores of abdominal pain (0-3), general well-being (0-4, higher values mean worse well-being), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome. Change from baseline in abdominal pain was reported.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 96, Week 156, Week 216, Week 264, and Week 300
Population: Participants from safety analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 911 | 113 | 113
units on a scale
  Baseline | 1.6 (0.91) | 1.0 (0.89) | 0.7 (0.75)
  Change at Week 12: number analyzed (Participants) | 787 | 103 | 103
  Change at Week 12 | -0.6 (0.91) | -0.2 (0.65) | 0.0 (0.52)
  Change at Week 24: number analyzed (Participants) | 682 | 89 | 89
  Change at Week 24 | -0.7 (0.92) | -0.2 (0.75) | 0.0 (0.51)
  Change at Week 48: number analyzed (Participants) | 516 | 74 | 81
  Change at Week 48 | -0.8 (0.97) | -0.3 (0.70) | -0.1 (0.54)
  Change at Week 96: number analyzed (Participants) | 305 | 49 | 53
  Change at Week 96 | -0.8 (1.00) | -0.2 (0.73) | 0.0 (0.55)
  Change at Week 156: number analyzed (Participants) | 117 | 30 | 26
  Change at Week 156 | -0.8 (0.98) | -0.2 (0.77) | 0.0 (0.57)
  Change at Week 216: number analyzed (Participants) | 82 | 13 | 6
  Change at Week 216 | -0.9 (1.05) | -0.5 (0.88) | 0.0 (0.00)
  Change at Week 264: number analyzed (Participants) | 20 | 4 | 0
  Change at Week 264 | -0.8 (0.64) | -1.3 (0.50) |
  Change at Week 300: number analyzed (Participants) | 4 | 0 | 0
  Change at Week 300 | -0.3 (0.50) |  |

4. Secondary Outcome: Change From Baseline in CDAI Scores
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The sub scores of abdominal pain (rated on a scale of 0-3, higher values mean greater abdominal pain), general well-being (0-4, higher values mean worse well-being), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
Time Frame: Baseline, Week 12, Week 24, Week 48, Week 96, Week 156, Week 216, Week 264, and Week 300
Population: Participants from safety analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 897 | 110 | 110
units on a scale
  Baseline | 280.5 (116.58) | 189.9 (112.73) | 120.4 (81.33)
  Change at Week 12: number analyzed (Participants) | 710 | 94 | 92
  Change at Week 12 | -86.8 (114.02) | -29.1 (79.84) | 4.2 (53.42)
  Change at Week 24: number analyzed (Participants) | 608 | 84 | 82
  Change at Week 24 | -98.5 (122.68) | -30.8 (92.92) | 5.7 (51.30)
  Change at Week 48: number analyzed (Participants) | 461 | 69 | 71
  Change at Week 48 | -110.2 (125.08) | -40.9 (91.47) | 0.6 (49.32)
  Change at Week 96: number analyzed (Participants) | 261 | 46 | 45
  Change at Week 96 | -118.6 (131.49) | -23.3 (91.94) | 11.0 (69.29)
  Change at Week 156: number analyzed (Participants) | 154 | 28 | 24
  Change at Week 156 | -121.4 (132.33) | -33.5 (99.15) | 0.3 (59.27)
  Change at Week 216: number analyzed (Participants) | 65 | 13 | 4
  Change at Week 216 | -137.0 (147.14) | -57.5 (121.12) | 2.5 (37.76)
  Change at Week 264: number analyzed (Participants) | 16 | 4 | 0
  Change at Week 264 | -134.8 (128.86) | -171.5 (141.81) |
  Change at Week 300: number analyzed (Participants) | 4 | 0 | 0
  Change at Week 300 | -32.5 (92.99) |  |

ADVERSE EVENTS:
Time Frame: From the First Dose to Week 312
Description: Safety Analysis Set
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 6/944 | 2/119 | 1/124
Serious Adverse Events (participants affected / at risk) | 284/944 | 34/119 | 20/124
Other Adverse Events (participants affected / at risk) | 697/944 | 89/119 | 78/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filgotinib 200 mg (N=944) | Filgotinib 100 mg (N=119) | Placebo (N=124)
Parathyroid tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cervix injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture of penis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 7 (11) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 17 (18) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dental necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 101 (108) | 5 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colon dysplasia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 8 (9) | 2 (2) | 0 (0)
Intestinal mucosal tear (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 2 (5) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 11 (14) | 9 (10) | 3 (3)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 15 (18) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis cryptosporidial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filgotinib 200 mg (N=944) | Filgotinib 100 mg (N=119) | Placebo (N=124)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (16) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 40 (41) | 8 (8) | 3 (3)
Pyrexia (General disorders) | 65 (94) | 3 (4) | 0 (0)
Fatigue (General disorders) | 35 (40) | 5 (6) | 4 (6)
Asthenia (General disorders) | 20 (24) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 24 (26) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 23 (24) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 20 (20) | 3 (3) | 1 (1)
Mycobacterium tuberculosis complex test positive (Investigations) | 12 (12) | 0 (0) | 5 (5)
Weight decreased (Investigations) | 22 (22) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4) | 3 (3) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 79 (95) | 4 (5) | 11 (12)
Dizziness (Nervous system disorders) | 26 (28) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 27 (34) | 2 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 22 (23) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 61 (73) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 21 (27) | 5 (5) | 5 (6)
Anal fistula (Gastrointestinal disorders) | 24 (31) | 3 (3) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 24 (27) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 93 (126) | 15 (19) | 15 (18)
Abdominal distension (Gastrointestinal disorders) | 17 (19) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 67 (86) | 3 (3) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 10 (12) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 74 (83) | 8 (8) | 4 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22 (24) | 3 (3) | 1 (1)
Gastritis (Gastrointestinal disorders) | 16 (16) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 29 (31) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 54 (66) | 10 (13) | 11 (12)
Crohn's disease (Gastrointestinal disorders) | 210 (269) | 26 (36) | 20 (22)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 27 (29) | 7 (7) | 2 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 11 (11) | 7 (9) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 (18) | 4 (4) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 43 (53) | 4 (5) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 (103) | 15 (24) | 1 (3)
Urinary tract infection (Infections and infestations) | 57 (82) | 8 (14) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 57 (84) | 8 (9) | 3 (4)
Sinusitis (Infections and infestations) | 30 (35) | 7 (9) | 0 (0)
Pharyngitis (Infections and infestations) | 18 (22) | 1 (1) | 3 (3)
Oral herpes (Infections and infestations) | 14 (19) | 3 (4) | 0 (0)
Anal abscess (Infections and infestations) | 16 (22) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 30 (37) | 5 (5) | 2 (4)
COVID-19 (Infections and infestations) | 127 (139) | 17 (17) | 9 (10)
Gastroenteritis (Infections and infestations) | 26 (29) | 4 (5) | 1 (1)
Herpes zoster (Infections and infestations) | 22 (22) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 27 (31) | 4 (5) | 4 (6)
Latent tuberculosis (Infections and infestations) | 14 (14) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 81 (101) | 13 (21) | 6 (6)
Folate deficiency (Metabolism and nutrition disorders) | 13 (14) | 3 (5) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (24) | 3 (4) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 30 (35) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 21 (23) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The results of DIVERSITY 1 study with filgotinib in participants with moderate to severely active CD failed to meet the co-primary endpoints of clinical remission and endoscopic response for filgotinib 100 mg q.d. and 200 mg q.d. in the study. After analyzing all available data from the DIVERSITY 1 and DIVERSITY long term extension (LTE) studies, the sponsor decided not to pursue extension of the filgotinib indication for CD and decided to terminate the DIVERSITY LTE study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02914600/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT02914600/SAP_001.pdf